CLINICAL TRIAL: NCT03071991
Title: Effect of Preincisional Bupivakain Infiltration on Postoperative Narcotic Medication in Laparoscopic Sleeve Gastrectomy
Brief Title: Effect of Preincisional Bupivakain Infiltration on Postoperative Narcotic Medication Requirement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdullah Sisik, General Surgery Specialist, Umraniye Education and Research Hospital
Other Study IDs: PREINS-BUP-POSTOP-NARCOTIC-REQ
Record Dates: First submitted 2017-01-05; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Pain, Postoperative
Keywords: preinsicional bupivacain; laparoscopic bariatric surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Study group: Preincisional bupivacain will be used
  Interventions: Procedure: study group
- Control group: No preincisional anesthetic drug will be used
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: study group — local anesthetic drug will be used
  Groups: Study group
Procedure: control group — no local anesthetic drug will be used
  Groups: Control group

SUMMARY:
Postoperative pain and use of narcotic analgesics after laparoscopic bariatric surgeries are problems that need to be solved in terms of patient comfort. We believe that preincisional bupivacain injection to the trocar sites will help us for these problems. A study is designed focused on reduced postoperative pain and reduced use of narcotic analgesics by preincisional bupivacain injection for laparoscopic bariatric patients.

DETAILED DESCRIPTION:
A randomised controlled prospective study is designed with 40 patients over 2-month period (January 2017 to february 2017). Laparoscopic sleeve gastrectomy is planned for all patients. Two groups are designed depending on whether trocar site infiltration with bupivacaine was performed (study group, 20 patients) or not (control group, 20 patients). The patients with body mass index (BMI) ≥35kg/m2 are enrolled to study. The parameters of demographic characteristics (age, gender, BMI, weight, and body fat percentage), preoperative comorbid conditions (type 2 diabetes mellitus, hypertension), and clinical outcomes (postoperative complications, mortality, readmissions) are planned to record.

Pain evaluation

Visual analogue scale (VAS, 0: no pain, 10: the worst imaginable pain) is planned to be used. VAS measurements timing is planned as follows:

* first postoperative day: 4th, 8th, 12th, and 24th hours
* second postoperative day: 48th hour.

Operative Technique

All patients will be operated by same surgeons and anesthetist. Peroperatively intravenous paracetamol 10 mg, tramadol 50 mg and fentanyl 150 mcg will be used for analgesia. Local infiltration of the port sites was carried out through out all layers with 40 ml 0.25% bupivacaine and 1:200,000 epinephrine before incision. Laparoscopic sleeve gastrectomy will be performed with 5 trocars, in reverse trandelenburg position by creating pneumoperitoneum with 14 mmHg carbon dioxide insufflation. Trocar replacements are one 10-mm trocar in the midline above umbilicus for the endoscope, one 12-mm trocar to right midclavicular line linage to the 10-mm trocar. One 5-mm trocar to the left midclavicular line linage to the 10-mm trocar, one 5-mm trocar to the front axiller line below the left costal margin, and 5-mm trocar 2 cm below the xiphoid process for liver retractor. 38 F orogastric tube will be used. No use of nasogastric tubes and urinary catheters routinely is planned. Drain replacement is planned for all patients.

Postoperative Management

All patients will be mobilised 4th postoperative hour, and all patients will use breathing exercise device hourly. Postoperative analgesia protocol is designed with intravenous paracetamol 1 g every 8 h and deksketoprofen trometamol 50 mg every 12 h, antiemetics (ondansetron 4 mg every 8 h). Narcotic analgesic pethidin hcl 50 mg/ml will be ordered to patients who had > 5 degrees of pain according to VAS. The patients are Oral liquid diet was started on the second postoperative day, advanced to semisolid diet after discharging.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for bariatric surgery

Exclusion Criteria:

* Refusal for participating to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with body mass index (BMI) ≥35kg/m2 will be enrolled to the study. Laparoscopic sleeve gastrectomy will be planned for study patients .
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | postoperative 48 hours
  VAS scale will be used
postoperative narcotic drug need | postoperative 48 hours
  VAS scale will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Nazif Bagriacik Kadikoy Hospital, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No